CLINICAL TRIAL: NCT01981811
Title: A Single-arm Study to Evaluate Adherence to Treatment With, and Safety and Tolerability of, the Medical Information Device #1 (MIND1) System in Subjects With Schizophrenia or Bipolar I Disorder Who Are Currently Treated With Oral Aripiprazole
Brief Title: Adherence to Treatment, Safety and Tolerability Study of the Medical Information Device #1 (MIND1) in Subjects With Schizophrenia or Bipolar I Disorder
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial was terminated because it was determined that the usability of the MIND1 System in the intended population was necessary before conducting this trial.
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 316-13-211
Record Dates: First submitted 2013-10-22; First posted 2013-11-13 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Bipolar 1 Disorder; Schizophrenia; Mental Disorder; Nervous System Diseases
Keywords: OPC-14597 Digital; Aripiprazole; Medical Information Device #1 System (MIND1); Treatment Adherence; Ingestible Event Marker
MeSH Terms: conditions — Schizophrenia; Mental Disorders; Nervous System Diseases; Treatment Adherence and Compliance | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aripiprazole and Ingestible Event Marker (IEM) (Active Comparator): All subjects will continue to receive their previously prescribed dose of aripiprazole (10 mg, 15 mg, 20 mg, or 30 mg) through the trial. Subjects will discontinue dosing of the conventional oral aripiprazole tablet and will begin taking MIND1 (aripiprazole embedded with an Ingestible Event Marker) tablet once-daily for 12 weeks.
  Interventions: Drug: Aripiprazole; Device: Ingestible Event Marker (IEM)

INTERVENTIONS:
Drug: Aripiprazole
Device: Ingestible Event Marker (IEM)

SUMMARY:
The purpose of this study is to evaluate adherence to treatment with, and safety and tolerability of, the medical information device #1 (MIND1) system in subjects with Schizophrenia or Bipolar I Disorder who are currently treated with oral aripiprazole.

DETAILED DESCRIPTION:
Poor adherence to medication is a well-recognized problem in psychiatric patients and is a barrier to achieving optimal health. The MIND1 System is being developed to objectively and precisely monitor and measure real-time medication adherence; and to potentially enhance adherence. The MIND1 System includes oral aripiprazole with an embedded ingestible event marker (IEM), a Wearable Sensor, and a computerized device and accessories. This is a trial designed to evaluate adherence to treatment with, and safety and tolerability of, the medical information device #1 (MIND1) system in subjects with schizophrenia or bipolar I disorder. This 12-week, single-arm trial will include male and female subjects 18 to 65years (inclusive) with a current diagnosis of schizophrenia or bipolar I disorder who are currently treated with oral aripiprazole.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 to 65 years of age, inclusive, at time of informed consent
* Schizophrenia: Patients with two or more exacerbations of symptoms in past year leading to an intervention, per investigator's judgment (ie, inpatient psychiatric hospitalization, psychiatric ER visit, admission to partial hospitalization program, crisis residential treatment, etc.). This does not include outpatient adjustment of medication.
* Bipolar I Disorder: Patients with at least one manic episode or exacerbation of bipolar symptoms in past year resulting in an intervention, per Investigator's judgment (i.e., inpatient psychiatric hospitalization, psychiatric ER visit, admission to partial hospitalization program, crisis residential treatment, etc.) This does not include outpatient adjustment of medication.
* Current primary Axis-1 diagnosis of bipolar 1 disorder or schizophrenia as defined by DSM-IV-TR criteria
* Bipolar 1 disorder patients with a total YMRS score of 10 to 25 (inclusive)
* Schizophrenia patients with a total PANSS score of 60 to 90 (inclusive)
* Currently prescribed oral Aripiprazole for either bipolar 1 disorder or schizophrenia. No changes in their Aripiprazole dose or regimen 2 weeks before screening.
* Subjects must be able to tolerate blood draws.
* If subject is on other psychotropic medications, he/she must be on a stable dose and regimen over the last 2 weeks.

Exclusion Criteria:

* Subjects with a current Axis I (DSM-IV-TR) diagnosis other than bipolar 1 disorder or schizophrenia
* Subjects with a current Axis II (DSM-IV-TR) diagnosis
* History of inpatient hospitalization for any psychiatric reason within 2 months before screening
* Subjects who reside or attend a facility where medication is administered to them
* Subject has received any investigational product within the last 30 days
* Allergic, intolerant, or unresponsive to prior treatment with Aripiprazole or other quinolinones
* History of hypersensitivity to antipsychotic agents

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2014-05 (Actual); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Medication adherence, as defined by the number of IEM detections reported by the MIND1 System divided by the medication doses prescribed. | Baseline to Week 12

SECONDARY OUTCOMES:
Compliance, defined as the ratio of individual model-predicted exposure (AUC) at Week 12 following administration of oral aripiprazole using the MIND1 System versus the expected exposure | Week 12

OTHER OUTCOMES:
Comparison of the predicted PK exposure (log transformed-area under the plasma concentration-time curve [AUC]) at Week 12 to the predicted PK exposure prior to use of the MIND1 System | Week 12
Change in compliance, defined as the difference in predicted adherence at Week 12 and the predicted adherence before using the MIND1 System | Week 12
Proportion of subjects who achieve greater than 80% compliance post-Week 12 administration of aripiprazole through MIND1 | Baseline to Week 12
Severity of illness, defined by the change from Screening/baseline to Week 12 with scores on the CGI-scale, PSP, SLOF, PANSS and YMRS. | Screening/baseline to Week 12
Safety and tolerability: frequency and severity of AEs; frequency of serious AEs; AEs leading to discontinuation; and frequency and severity of unexpected adverse events and unanticipated device adverse events (UDAE) | Baseline to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Shashank Rohatagi, PhD, Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (12):
- United States (12):
  - Cerritos, California
  - Garden Grove, California
  - Long Beach, California
  - National City, California
  - Oceanside, California
  - San Diego, California
  - Washington D.C., District of Columbia
  - Atlanta, Georgia
  - St Louis, Missouri
  - Marlton, New Jersey
  - Dayton, Ohio
  - Irving, Texas